CLINICAL TRIAL: NCT03194022
Title: Per Effort Study of Biological Consequences of an Ultra Endurance Race (165km)
Brief Title: Biological Consequences of an Ultra Endurance Race
Acronym: TRAIL-BIO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Principal Investigator, Romain Jouffroy, Principal Investigator, Hôpital Necker-Enfants Malades
Other Study IDs: IDRCB : 2017-A01801-52
Record Dates: First submitted 2017-06-16; First posted 2017-06-21 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Exertion; Excess
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood electrolytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sample — measurement of electrolytes and blood count

SUMMARY:
The aim is to study per and post-exertion variations of biological markers during an ultra-endurance race

DETAILED DESCRIPTION:
25 healthy adult volunteers participating in the "100 miles South of France 2017©" race recruited electronically by an announcement on the race website

ELIGIBILITY:
Inclusion Criteria:

1. Age greater 18 years.
2. Subject having already completed an ultra-endurance race (distance greater than 50 kilometers) during the 24 months preceding the race.
3. Affiliation of a social security.

Exclusion Criteria:

1. Age lower than 18 years
2. Subjects with a medical history (pulmonary pathology, cardiac, hypertension) or having a significant chronic inflammatory disease known at the time of the inclusion visit the day before the race.
3. Female

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 healthy adult volunteers participating in the "100 miles South of France 2017 ©" race recruited electronically by an announcement on the race website
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-17 (Estimated)

PRIMARY OUTCOMES:
Per and post-exertion evolution of sodium blood level | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  Change of sodium blood level during and after the race will be measured.
Per and post-exertion evolution of lactatemia | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  Change of lactatemia during and after the race will be measured.
Per and post-exertion evolution of myoglobin blood level | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  Change of myoglobin blood level will be measured during and after the race
Per and post-exertion evolution of creatinine phosphokinase blood level | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  Change of myoglobin blood level will be measured during and after the race
Per and post-exertion evolution of potassium blood level | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  Change of potassium blood level during and after the race will be measured.
Per and post-exertion evolution of chlorine blood level | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  Change of chlorine blood level during and after the race will be measured.
Per and post-exertion evolution of glucose blood level | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  Change of glucose blood level during and after the race will be measured.
Per and post-exertion evolution of calcium blood level | Change measures : departure, 15, 50, 65, 90, 130 and 165 kilometers then at day 1 and 2 after the completion of the race
  Change of calcium blood level during and after the race will be measured.

IPD SHARING:
Plan to Share IPD: Undecided